CLINICAL TRIAL: NCT07107607
Title: Cannabis as an Anti-cancer Agent: A Review of Medical Records in Patients With Cancer to Assess Potential Anti-cancer Benefits From Using Cannabis
Brief Title: Assessing Claims of Cannabis as an Anti-cancer Agent (CATA)
Acronym: CATA
Status: Recruiting | Type: Observational
Sponsor: HealthPartners Institute (Other)
Responsible Party: Sponsor
Other Study IDs: CATA
Record Dates: First submitted 2025-07-25; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Cancer; Cancer (With or Without Metastasis)
Keywords: cancer; cannabis; marijuana; tetrahydrocannabinol; cannabidiol
MeSH Terms: conditions — Neoplasms; Marijuana Abuse

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the study is to find out how cannabis may help control cancer growth by reviewing medical records of patients who report cannabis helped treat their cancer.

DETAILED DESCRIPTION:
The purpose of the study is to further assess how cannabis may help control cancer growth and attempt to validate such claims. To do this, the investigators will review medical records from consented patients who report that cannabis has helped to reduce or control growth of cancer by assessing prior cancer treatments and assessments (for example, cancer/tumor labs like prostate-specific antigen (PSA), cancer antigen (CA)-125, carcinoembryonic antigen (CEA) and radiology imaging reports such as computed tomography (CT) scan, positron emission tomography (PET)/CT scan, and magnetic resonance imaging (MRI)) as well as cannabis use details.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with cancer
* have used any type of cannabis/marijuana, including those with cannabidiol (CBD) and/or tetrahydrocannabinol (THC) to treat their cancer
* believe that cannabis has either stopped the tumor from growing and/or caused a cancer antigen blood marker to remain stable or cannabis has shrunken the tumor and/or caused reduction in a cancer antigen blood marker

Exclusion Criteria:

* does not have cancer
* has not used any type of cannabis/marijuana, including those with CBD and/or THC to treat their cancer
* does not believe that cannabis has either stopped the tumor from growing and/or caused a cancer antigen blood marker to remain stable or cannabis has shrunken the tumor and/or caused reduction in a cancer antigen blood marker

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: people with cancer who report that cannabis use had an impact on their cancer growth
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-03-19 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
To successfully complete Phase 2 by recruiting patients to consent with a simplified screening survey. | From enrollment start to the obtainment of cancer diagnosis and treatment details and cannabis use history from each consented patient, which is estimated to take up to 6 years.
  Successful completion of phase 2 of this survey study will include consenting 50 patients and obtaining their cancer and cannabis use details to validate anti-cancer claims.

CONTACTS AND LOCATIONS:
Locations (1):
- HealthPartners Institute Cancer Research Center, Saint Louis Park, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No